CLINICAL TRIAL: NCT01981967
Title: Post-licensure, Phase IV, Safety Study of IMOJEV® in Thailand
Brief Title: Post-licensure Safety Study of IMOJEV® in Thailand
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JEC17; U1111-1127-7052 (Other: WHO)
Record Dates: First submitted 2013-11-05; First posted 2013-11-13 (Estimated); Results first posted 2016-05-04 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-03

CONDITIONS: Japanese Encephalitis
Keywords: Japanese encephalitis; IMOJEV®; Japanese encephalitis chimeric virus vaccine
MeSH Terms: conditions — Encephalitis, Japanese

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Primary Vaccination Group (Experimental): Participants who never received a JE vaccine, or who received a single dose of inactivated JE vaccine, or whose JE vaccination history is unknown or not documented.
  Interventions: Biological: IMOJEV®: Live attenuated Japanese encephalitis chimeric virus vaccine
- Booster Vaccination Group (Active Comparator): Participants who received at least 2 doses of inactivated JE vaccine (at least 1 year earlier for the last dose), or received a single dose of IMOJEV®, THAIJEV®, or IMOJEV® MD as part of the routine vaccination schedule (i.e., outside of Study JEC17) at least 1 year earlier
  Interventions: Biological: IMOJEV®: Live attenuated Japanese encephalitis chimeric virus vaccine

INTERVENTIONS:
Biological: IMOJEV®: Live attenuated Japanese encephalitis chimeric virus vaccine — 0.5 mL, Subcutaneous.
  Other Names: IMOJEV®
  Arms: Primary Vaccination Group
Biological: IMOJEV®: Live attenuated Japanese encephalitis chimeric virus vaccine — 0.5 mL, Subcutaneous.
  Other Names: IMOJEV®
  Arms: Booster Vaccination Group

SUMMARY:
The aim of this study is to further characterize the safety profile of IMOJEV®.

Primary Objective:

* To describe serious adverse events (SAEs, including adverse events of special interest [AESIs]) up to 60 days after administration of one dose of IMOJEV®.

Secondary Objective:

* To describe Grade 3 (severe) systemic Adverse Events (AEs) up to 30 minutes after administration of one dose of IMOJEV®.

DETAILED DESCRIPTION:
Participants aged 1 year to less than 5 years will be randomized to receive one injection of IMOJEV® either as a primary vaccination or as a booster. Safety data will be collected for 60 days after IMOJEV® vaccination. The duration of each subject's participation in the trial will be 60 days.

ELIGIBILITY:
Inclusion Criteria:

* Children requiring vaccination against Japanese encephalitis
* Children aged 9 months to less than 5 years on the day of inclusion
* In good general health at the time of inclusion
* Informed consent form has been signed and dated by the parent(s)/legal guardian(s)
* Subject and parent(s)/legal guardian(s) are able to attend the scheduled visit and any additional visits that may need to be done in case of an SAE (including AESI), and are able to comply with all trial procedures
* The subject's parent(s)/legal guardian(s) have a telephone number at which they can be contacted throughout the study

Exclusion Criteria:

* Participation in another clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the vaccination
* Receipt of any vaccine in the 4 weeks preceding the study vaccination or planned receipt of any vaccine in the 4 weeks following the study vaccination
* Planned participation in another clinical trial during the present trial period
* Children previously vaccinated with the live attenuated Japanese encephalitis vaccine CD-JEVAX® (SA14-14-2 LAV)
* Contraindications to vaccination according to the IMOJEV® Summary of Product Characteristics (SmPC)
* Identified as a natural or adopted child of the Investigator or employee with direct involvement in the proposed study
* Children who received IMOJEV® as primary vaccination in this study.

Ages: 9 Months to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10000 (Actual)
Dates: Start 2013-11; Primary Completion 2015-04 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (7):
- Thailand (7):
  - Bangkok
  - Chiang Mai
  - Khon Kaen
  - Nakornnayok
  - Nonthaburi
  - Pathum Thani
  - Songkhla

REFERENCES:
- [Derived] Chotpitayasunondh T, Pruekprasert P, Puthanakit T, Pancharoen C, Tangsathapornpong A, Oberdorfer P, Kosalaraksa P, Prommalikit O, Tangkittithaworn S, Kerdpanich P, Techasaensiri C, Korejwo J, Chuenkitmongkol S, Houillon G. Post-licensure, phase IV, safety study of a live attenuated Japanese encephalitis recombinant vaccine in children in Thailand. Vaccine. 2017 Jan 5;35(2):299-304. doi: 10.1016/j.vaccine.2016.11.062. Epub 2016 Nov 28. PMID 27903416
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study participants were enrolled from 03 November 2013 to 08 February 2015 in 10 trial centers in Thailand.
Pre-assignment Details: A total of 10,000 participants who met all of the inclusion and none of the exclusion criteria were vaccinated in this study.
Groups:
- Primary Vaccination Group: Children aged 9 months to less than 5 years who received one injection of IMOJEV® as a primary vaccination.
- Booster Vaccination Group: Children aged 9 months to less than 5 years who received one injection of IMOJEV® as a booster.
Period: Overall Study
Arm/Group | Primary Vaccination Group | Booster Vaccination Group
Started | 6851 | 3149
Completed | 6851 | 3149
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Primary Vaccination Group | Booster Vaccination Group | Total
Number analyzed (Participants) | 6851 | 3149 | 10000
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6851 | 3149 | 10000
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 1.22 (0.486) | 3.60 (0.892) | 1.97 (1.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3321 | 1550 | 4871
  Male | 3530 | 1599 | 5129
Region of Enrollment [Number; unit: Participants]
  Thailand | 6851 | 3149 | 10000

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing a Grade 3 Immediate Systemic Adverse Events and Serious Adverse Events Following Any Vaccination With IMOJEV®
Time Frame: 30 minutes post-vaccination up to Day 60 post-vaccination
Population: Safety outcome were assessed in subjects who had received the study vaccine, the Safety Analysis Set
Measure: Number; unit: Participants
Arm/Group | Primary Vaccination Group | Booster Vaccination Group
Number analyzed (Participants) | 6851 | 3149
Participants
  Grade 3 immediate systemic adverse event | 0 | 0
  Seriuos adverse events | 204 | 59
  Death | 0 | 1

2. Primary Outcome: Number of Participants Experiencing Serious Adverse Events By Age Following Any Vaccination With IMOJEV®
Time Frame: Day O up to Day 60 post-vaccination
Population: Safety outcome were assessed in subjects who had received the study vaccine, the Safety Analysis Set
Measure: Number; unit: Participants
Arm/Group | Primary Vaccination Group | Booster Vaccination Group
Number analyzed (Participants) | 6851 | 3149
Participants
  SAEs in Subjects 9 to <12 Months | 43 | 0
  SAEs in Subjects 1 to 2 Years | 155 | 0
  SAEs in Subjects 2 to <5 Years | 6 | 59

3. Secondary Outcome: Number of Participants Experiencing Adverse Events of Special Interest Within 60 Days Following Vaccination With IMOJEV®
Description: Adverse Events of Special Interest (AESIs) included hypersensitivity/allergic reactions, neurological events (including febrile convulsions), and vaccine failure.
Time Frame: Day O up to Day 60 post-vaccination
Population: Safety outcome were assessed in subjects who had received the study vaccine, the Safety Analysis Set
Measure: Number; unit: Participants
Arm/Group | Primary Vaccination Group | Booster Vaccination Group
Number analyzed (Participants) | 6851 | 3149
Participants
  Febrile convulsion | 25 | 2
  Convulsion | 1 | 0
  Epilepsy | 1 | 0
  Frontal lobe epilepsy | 1 | 0
  Urticaria | 0 | 2

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 (post-vaccination) up to 60 post-vaccination
Arm/Group | Primary Vaccination Group | Booster Vaccination Group
Serious Adverse Events (participants affected / at risk) | 204/6851 | 59/3149
Other Adverse Events (participants affected / at risk) | 0/6851 | 0/3149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary Vaccination Group (N=6851) | Booster Vaccination Group (N=3149)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 8 (8) | 4 (4)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Allergy to arthropod sting (Immune system disorders) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Acute tonsillitis (Infections and infestations) | 4 (4) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 6 (6) | 0 (0)
Bronchitis (Infections and infestations) | 17 (17) | 10 (10)
Bronchitis viral (Infections and infestations) | 1 (1) | 0 (0)
Burkholderia pseudomallei infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Croup infectious (Infections and infestations) | 2 (2) | 0 (0)
Dengue fever (Infections and infestations) | 1 (1) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 5 (5) | 0 (0)
Exanthema subitum (Infections and infestations) | 1 (1) | 0 (0)
Gastritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 28 (29) | 8 (8)
Gastroenteritis rotavirus (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 4 (4) | 0 (0)
Hand-foot-mouth disease (Infections and infestations) | 6 (6) | 2 (2)
Herpangina (Infections and infestations) | 1 (1) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 1 (1) | 2 (2)
Influenza (Infections and infestations) | 4 (4) | 5 (5)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 3 (3)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Otitis media acute (Infections and infestations) | 3 (3) | 0 (0)
Pharyngitis (Infections and infestations) | 10 (10) | 0 (0)
Pharyngitis bacterial (Infections and infestations) | 2 (2) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 24 (24) | 7 (7)
Pneumonia bacterial (Infections and infestations) | 4 (4) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 4 (4) | 0 (0)
Pneumonia viral (Infections and infestations) | 10 (11) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 (1) | 1 (1)
Respiratory syncytial virus bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Scarlet fever (Infections and infestations) | 1 (1) | 0 (0)
Scrotal abcess (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 1 (1)
Urinary track infection (Infections and infestations) | 6 (6) | 0 (0)
Viral diarrhoea (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 2 (2) | 0 (0)
Viral rash (Infections and infestations) | 2 (2) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Febrile convulsion (Nervous system disorders) | 25 (28) | 2 (2)
Frontal lobe epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Kawasaki's disease (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications